CLINICAL TRIAL: NCT06374927
Title: Personalised Health Cognitive Assistance for RehAbilitation SystEm (PHRASE): A Feasibility Study
Acronym: PHRASE-2023
Status: Recruiting | Type: Observational
Sponsor: Donders Centre for Neuroscience (Other)
Responsible Party: Principal Investigator, Paul Verschure, Responsible Party, Donders Centre for Neuroscience
Other Study IDs: PHRASE-2023
Record Dates: First submitted 2024-04-16; First posted 2024-04-19 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Stroke
Keywords: Stroke; Rehabilitation; Virtual Reality (VR); Augmented Reality (AR)
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Stroke patients: Stroke patients at different time points after stroke (acute, subacute, and chronic), aged over 18 years.
  Interventions: Device: Rehabilitation Gaming System (VR-based mobile application)

INTERVENTIONS:
Device: Rehabilitation Gaming System (VR-based mobile application) — The study intervention includes using the mobile phone technology RGSapp. This application integrates sensor data for delivering patient-tailored VR and AR-based training via gamified exercises for cognitive training.

SUMMARY:
The incidence of cognitive and neuromotor impairment caused by strokes has become a growing challenge.

The patient's journey to recovery in the healthcare system involves multiple phases, spanning from initial hospitalization to in-patient and out-patient rehabilitation, finally leading to the patient's return to home. The access to stroke units and rehabilitation varies within Europe. Unfortunately, not everyone has access to rehabilitation programs, and the benefits derived from these programs often decline after hospital discharge.

Currently, the support of the patient is organized in a rather fragmented way, and informal care sometimes places a severe burden requiring dedicated support in the patient's social environment. The PHRASE project proposes to deploy rehabilitation technology such as the Rehabilitation Gaming System (RGS) to instil and support a virtuous cycle of stroke patients' recovery in the at-home setting. RGS is an effective advanced digital tool for rehabilitation programs that uses Augmented Reality (AR)- and Virtual Reality (VR)-based gamified training grounded on neuroscientiﬁc principles, that has been shown to promote cognitive and motor recovery after a stroke at the clinic and home.

There are many dedicated cognitive therapies, but most rehabilitation outcomes are mostly limited to the task trained and do not extend to day-to-day function or remain unconvincing. Based on recent literature, the PHRASE RGS-based system can provide an effective tool to address cognitive impairment using VR-based interventions. In a previous study, the neuropsychological test battery was compiled by the neuropsychologist and covered four cognitive domains: 1. basic attention, 2. memory (short-term memory), 3. visuospatial memory, and 4. executive function. All these functions were tested using VR-based tasks. The conclusion of this study confirms the possibility of addressing cognitive impairment effectively using VR-based interventions when properly mapped with clinical scales.

The validation of the PHRASE system with post-stroke patients is needed to strengthen its usefulness and effectiveness for cognitive rehabilitation at home. For this, a feasibility study will be conducted to measure its usability, adherence, acceptance, and the user's experience.

The investigators will also explore the effectiveness of the PHRASE system in improving cognitive function (attention, memory, executive function) after stroke.

Participants: stroke patients at different time points after stroke (acute, subacute, and chronic), aged over 18 years. The participants will integrate the PHRASE technology into their daily routines in parallel to their regular neurorehabilitation treatment for 6 weeks.

DETAILED DESCRIPTION:
The rapid growth in the number of stroke patients needing care and rehabilitation requires an urgent scientifically grounded, and scalable response. There are many dedicated cognitive therapies, but most rehabilitation outcomes are mostly limited to the task trained and do not extend to day-to-day function or remain unconvincing. The PHRASE project combines theoretical neuroscience, and intervention protocols based on VR AR technology, the RGS, making it an excellent alternative to solving cognitive training.

The study is a feasibility study based on both quantitative and qualitative data collection. The general objective is to measure the usability of the system, including the user experience, adherence, and acceptance of the PHRASE system.

Specifically, the patient interacts with the RGSapp, a mobile app system that through the mobile registers the patient's movements and performance during the tasks to evaluate, reassess and update training protocols through AI-based algorithms. The clinicians have access to MIMS (Medical Information Management System) a portal that allows them to manage the patient profiles and deliver precise and objective metrics of the performance of the patient together with dashboards for therapists and clinicians. It facilitates diagnostics, monitoring, intervention scheduling, data storage and analytics, and reports and patient management.

The primary objective of this study is to measure the usability, adherence, user experience and acceptance of the PHRASE system during a six-week intervention.

Secondary outcome parameters will be assessed with clinical scales to explore the effectiveness of performing motor and cognitive assessments online and cognitive treatments provided through the RGSapp technology.

Investigators hypothesize that the personalized training supported by the PHRASE system is:

1. Highly accepted by patients and clinicians. More specifically, it is expected that this approach to show good user experience and usability by the patients and ease patients' management by the clinicians.
2. It increases the frequency and time spent with the rehabilitation program. More specifically, it is expected this approach shows good adherence to treatment.
3. Explore the impact of the PHRASE system on cognitive assessment, function impairment, and quality of life.

STUDY DESIGN AND POPULATION: The study is a feasibility study based on both quantitative and qualitative data collection. The general objective is to measure the usability of the system, the user experience, the adherence, and the acceptance of the PHRASE system. Each clinical site will include 30-50 stroke patients (in any stroke stage), minimum age of 18 years. Over six weeks, the participants will integrate the PHRASE system into their daily routines, running parallel to their regular neurorehabilitation treatment.

STUDY SETTING: The study will be conducted in parallel in different European hospitals. The experimentation involves 3 different phases: Baseline assessment (T0) before the start of the trial, remote assessment (T1) and Final evaluation (T2) at the end of the trial, after 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Patients presenting an ischemic or intracerebral haemorrhagic stroke
2. Age > 18 years old
3. Moderate to mild proximal upper limb motor impairment Medical Research Council Scale (MRC≥2).
4. Lesion localisation by clinical symptoms/signs.
5. Able to sit on a chair or a wheelchair to interact with the RGS system.
6. Minimal experience with smartphone technology based on the clinician's opinion
7. Willing to participate and agree to comply with the trial scheme and procedures
8. Must sign an Informed Consent Form (ICF) indicating that they understand the purpose and the procedures of the study.

Exclusion Criteria:

1. Presence of a condition or abnormality that, in the opinion of the investigator, would compromise the safety of the patient or the quality of the data.
2. Severe cognitive capabilities that prevent the execution of the experiment, either evaluated by the MoCA < 19 or based on the clinician's opinion.
3. Arteriovenous malformation or lesions not related to a stroke.
4. Severe associated impairments such as proximal but not distal spasticity, communication disabilities (sensory, Wernicke aphasia, or apraxia), major pain, or other neuromuscular impairments.
5. Pre-stroke history of upper limb motor disability.
6. Unable to use the RGS independently according to the clinician's observations and lacking support from a caregiver to use the RGS.
7. Refusal to sign the consent form.
8. No experience with smartphone technology or based on the clinician's opinion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Stroke patients at different time points after stroke (acute, subacute, and chronic).
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2024-04-25 (Estimated); Primary Completion 2024-10-01 (Estimated); Study Completion 2024-10-30 (Estimated)

PRIMARY OUTCOMES:
Usability | Week 6
  Usability will be assessed at T2 by the System Usability Scale (SUS): The System Usability Scale is a reliable tool for measuring usability. It consists of a 10-item questionnaire with five response options for respondents, from 'Strongly agree' to 'Strongly disagree'.
User experience | Week 6
  User experience will be assessed at T2 by the User Experience Questionnaire (UEQ): the scales of the questionnaire cover a comprehensive impression of user experience. Both classical usability aspects (efficiency, perspicuity, dependability) and user experience aspects (originality, stimulation) are measured.
Adherence | Week 6
  Adherence will be assessed by the total time the RGSapp is used, in comparison to the advised RGSapp sessions for the entire duration of the study. Via the user ID, it is possible to monitor the patient's access to the RGSapp and the hours trained.
Acceptance | Week 6
  Acceptance will be assessed at T2 by Quebec User Evaluation of Satisfaction with Assistive Technology (QUEST 2.0): the instrument is a self-administered questionnaire assessing user satisfaction with assistive technology products and associated services.

SECONDARY OUTCOMES:
The Montreal Cognitive Assessment (MoCA) | Baseline, Week 6
  MoCA is a cognitive test validated as a highly sensitive tool for early detection of mild cognitive impairment (MCI). MoCA accurately and quickly assess the following: short-term memory, visuospatial abilities, executive functions, attention, concentration and working memory, language and orientation to time and place.
Fugl-Meyer Assessment of the sensorimotor function of the upper limb (FMA-UE) | Baseline, Week 6
  It is a stroke-specific and performance-based impairment index. It is designed to assess motor functioning, sensation, balance, and joint range of motion and joint pain in patients with post-stroke hemiplegia.
Hamilton Depression Rating Scale (HDRS) | Baseline, Week 6
  It is an instrument used for assessing symptoms of depression. It has been used in many key studies of depression and its treatment. The instrument is designed to be administered by clinicians after a structured or unstructured interview of the patient to determine their symptoms.
Fatigue Severity Scale (FSS) | Baseline, Week 6
  The Fatigue Severity Scale (FSS) is a nine-item unidimensional questionnaire designed to measure fatigue in people with chronic diseases. The scale is a self-report, paper-and-pencil requiring 2-3 min to be completed.
Pain Visual Analogue Scale (VAS) | Baseline, Week 6
  It is a one-dimensional measure of pain intensity used to record patients' pain progression. It is a horizontal/vertical straight line of fixed length, (100 mm), beginning and ending with the extreme limits of the evaluated parameter, oriented from left (worst) to right (best).
Barthel Index (BI) | Baseline, Week 6
  The Barthel Index is a measure of functional disability that assesses independence, mobility and the need for assistance in performing 10 common activities of daily living. Administration of the BI requires no special training or equipment.
EuroQol - 5 Dimension - 5 Level (EQ-5D-5L) | Baseline, Week 6
  The EuroQol - 5 Dimension - 5 Level (EQ-5D-5L): is a self-report survey that measures the quality of life across 5 domains: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension is scored on a 5-level severity ranking that ranges from 'No problems' through 'Extreme problems'.
Modified Ashworth scale (MAS) | Baseline, Week 6
  It is a muscle tone assessment scale that measures resistance during passive soft-tissue stretching.
  It is used as a simple measure of spasticity in patients with lesions of the Central Nervous System, it does not require any instrumentation and is quick to perform.

CONTACTS AND LOCATIONS:
Locations (4):
- Centre hospitalier universitaire de Limoges, Limoges, France
- Cluj Rehabilitation Hospital, Cluj-Napoca, Cluj, Romania
- Spain (2):
  - Parc Sanitari Sant Joan de Déu, Barcelona
  - IRF La Salle, Madrid